CLINICAL TRIAL: NCT01073969
Title: A Double-blind, Randomized, Controlled Crossover Trial to Assess the Digestive and Physiological Effects of a Wheat Bran Extract in Healthy Men and Women
Brief Title: Study to Determine the Digestive and Physiological Effects of an Extract From Bran in Healthy Men and Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kellogg Company (Industry)
Collaborators: Provident Clinical Research (Other); Tufts University (Other); University of Toronto (Other); University of Reading (Other); University of Saskatchewan (Other)
Responsible Party: Robin Dickmann, Senior Nutrition Scientist, Kellogg Company
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRV-08011
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: prebiotic study; modulating colonic bacteria
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control cereal (Placebo Comparator): grain-based ready to eat cereal that does not contain active wheat bran extract
  Interventions: Other: control wheat bran extract
- low dose (Active Comparator): grain-based ready to eat cereal containing a low dose of wheat bran extract
  Interventions: Other: wheat bran extract
- High dose (Active Comparator): grain-based ready to eat cereal that contains a high dose of wheat bran extract
  Interventions: Other: wheat bran extract

INTERVENTIONS:
Other: wheat bran extract — Comparison of control cereal (containing no added wheat bran extract)to two test cereals containing different amounts of added wheat bran extract
  Other Names: wheat bran oligosccharides; prebiotic oligosccharides
  Arms: High dose; low dose
Other: control wheat bran extract — Comparison of control cereal (containing no added wheat bran extract) to two test cereals containing different amounts of added wheat bran extract
  Other Names: wheat bran oligosccharides; prebiotic oligosccharides
  Arms: Control cereal

SUMMARY:
The primary objective of this trial is to determine whether two doses of an extract from bran demonstrate a prebiotic effect on colonic bacteria (by modulating selected fecal microbial populations, particularly bifidobacteria). The secondary objective is to measure the potential beneficial effects of consuming an extract from bran on the following physiological parameters: laxation, fecal pH, fecal moisture and stool consistency, blood glucose and insulin concentrations, plasma lipid profiles and serum free fatty acids, colonic bacterial short chain fatty acid production, ammonia metabolism and protein degradation, and biomarkers of oxidative stress and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18-75 years of age
* Body mass index ≥18.5 and <35.0 kg/m2
* Fasting LDL-C level ≥100 mg/dL and <200 mg/dL
* Otherwise judged to be in good health, willing to maintain habitual food and beverage intake and physical activity patterns throughout the trial

Exclusion Criteria:

* Significant gastrointestinal condition
* Use of pre/probiotic foods or supplements
* Use of antibiotics
* Pregnancy
* Certain muscle, liver, kidney, lung or gastrointestinal conditions and medications
* Poorly controlled hypertension
* Cancer treated within prior 2 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable will be the difference between treatments in bifidobacteria counts per g of feces, expressed as log10 cells per g feces (dry weight) | Baseline to end of each treatment (week 0 to week 3 of each treatment)

SECONDARY OUTCOMES:
Other fecal bacterial counts | baseline to end of each treatment (week 0 to week 3 of each treatment)
laxation | baseline to end of each treatment (week 0 to week 3 of each treatment)
fecal pH | baseline to end of each treatment (week 0 to week 3 of each treatment)
fecal moisture | baseline to end of each treatment (week 0 to week 3 of each treatment)
stool consistency | baseline to end of each treatment (week 0 to week 3 of each treatment)
blood glucose | baseline to end of each treatment (week 0 to week 3 of each treatment)
Blood insulin | baseline to end of each treatment (week 0 to week 3 of each treatment)
plasma lipid profiles | baseline to end of each treatment (week 0 to week 3 of each treatment)
serum free fatty acids | baseline to end of each treatment (week 0 to week 3 of each treatment)
fecal short chain fatty acids | baseline to end of each treatment (week 0 to week 3 of each treatment)
fecal ammonia | baseline to end of each treament (week 0 to week 3 of each treatment)
urinary para-cresol | baseline to end of each treatment (week 0 to week 3 of each treatment)
urinary phenol (total) | baseline to end of each treatment (week 0 to week 3 of each treatment)
urinary isoprostanes | baseline to end of each treatment (week 0 to week 3 of each treatment)
oxidized low density lipoprotein (TBARS, conjugated dienes) | baseline to end of each treatment (week 0 to week 3 of each treatment)
Urinary F2alpha-isoprostanes | baseline to end of each treatment (week 0 to week 3 of each treatment)
Plasma antioxidant capacity (ORAC, FRAP) | baseline to end of each treatment (week 0 to week 3 of each treatment)
serum amyloid A | baseline to end of each treatment (week 0 to week 3 of each treatment)
hs-CRP | baseline to end of each treatment (week 0 to week 3 of each treatment)
IL-6 | baseline to end of each treatment (week 0 to week 3 of each treatment)
TNF-alpha | baseline to end of each treatment (week 0 to week 3 of each treatment)
gastrointestinal symptom survey | baseline to end of each treatment (week 0 to week 3 of each treatment)
stool consistency (Bristol stool scale) | baseline to end of each treatment (week 0 to week 3 of each treatment)
Quality of Life questionaire (Quality Metrics SF-36) | baseline to end of each treatment (week 0 to week 3 of each treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, PhD, Study Director — Provident Clinical Research and Consulting, Inc
Locations (1):
- Provident CRC, Glen Ellyn, Illinois, United States